CLINICAL TRIAL: NCT05934955
Title: Safety, Tolerability, and Pharmacokinetics of Single Rising Oral Doses of BI 1839100 in Healthy Male Subjects (Single-blind, Randomised, Placebo-controlled, Parallel Group Design)
Brief Title: A Study in Healthy Men to Test How Well Different Doses of BI 1839100 Are Tolerated (1490-0003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1490-0003
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BI 1839100 low dose (Experimental)
  Interventions: Drug: BI 1839100
- BI 1839100 medium dose (Experimental)
  Interventions: Drug: BI 1839100
- BI 1839100 high dose (Experimental)
  Interventions: Drug: BI 1839100
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo matching BI 1839100

INTERVENTIONS:
Drug: BI 1839100 — BI 1839100
  Arms: BI 1839100 high dose; BI 1839100 low dose; BI 1839100 medium dose
Drug: Placebo matching BI 1839100 — Placebo matching BI 1839100
  Arms: Placebo

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability and pharmacokinetics (PK) of BI 1839100 in healthy male subjects following oral administration of single rising doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Japanese ethnicity, according to the following criteria: born in Japan, have lived outside of Japan <10 years, and have parents and grandparents who are Japanese
* Age of 18 to 45 years (inclusive)
* Body mass index (BMI) of 18.5 to 25 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Subjects who agree to minimise the risk of making their partner pregnant by fulfilling any of the following criteria starting from the start of trial medication until 90 days after end of trial medication:

  * Use of adequate contraception, any of the following methods plus condom: intrauterine device, combined oral contraceptives that started at least 2 months prior to the first drug administration
  * Vasectomized (vasectomy at least 1 year prior to enrolment)
  * Surgical sterilization (including bilateral tubal occlusion, hysterectomy or bilateral oophorectomy) of the subject's female partner

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre(s) of mercury (mmHg), diastolic blood pressure outside the range of 40 to 99 mmHg, or pulse rate outside the range of 40 to 99 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of any treatment-emergent adverse event assessed as drug-related by the investigator | up to 10 days

SECONDARY OUTCOMES:
Area under the concentration-time curve of plasma BI 1839100 over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 4 days
Maximum measured concentration of BI 1839100 in plasma (Cmax) | up to 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- SOUSEIKAI Sumida Hospital, Tokyo, Sumida-ku, Japan

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com